CLINICAL TRIAL: NCT01517776
Title: Cilengitide and Metronomic Temozolomide for Relapsed or Refractory High Grade Gliomas or Diffuse Intrinsic Pontine Gliomas in Children and Adolescents - A Phase II Study HIT-HGG-CilMetro - A Clinical Phase II Trial of the HIT-HGG Study Group -
Brief Title: Cilengitide and Metronomic Temozolomide for Relapsed or Refractory High Grade Gliomas or Diffuse Intrinsic Pontine Gliomas in Children and Adolescents
Acronym: HGG-CilMetro
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to an altered benefit/risk assessment.
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Principal Investigator, Christof Kramm, Principal investigator (, Martin-Luther-Universität Halle-Wittenberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIT-HGG-CilMetro; 2009-011898-33 (EudraCT Number)
Record Dates: First submitted 2012-01-11; First posted 2012-01-25 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-06

CONDITIONS: Gliomas
Keywords: High grade glioma; Glioblastoma multiforme; Anaplastic astrocytoma; Diffuse intrinsic pontine glioma; Relapse; refractory tumour disease; Relapsed or refractory high grade gliomas and diffuse intrinsic pontine gliomas
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma; Diffuse Intrinsic Pontine Glioma; Recurrence | interventions — Cilengitide; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cilengitide and metronomic temozolomide (Experimental): Cilengitide 1800 mg/m² i.v. twice weekly and Temozolomide 75 mg/m²/d p.o. for 6 weeks, followed by 1 week rest with a mandatory platelet-count dependent dose adaptation rule
  Interventions: Drug: Cilengitide; Drug: Temozolomide

INTERVENTIONS:
Drug: Cilengitide — Cilengitide 1800 mg/m² i.v. twice weekly with a mandatory platelet-count dependent dose adaptation rule
  Other Names: EMD 121974
Drug: Temozolomide — Temozolomide 75 mg/m²/d p.o. for 6 weeks, followed by 1 week rest with a mandatory platelet-count dependent dose adaptation rule
  Other Names: Temodal

SUMMARY:
The primary objective of this study is to evaluate the efficacy of a combined treatment with cilengitide and metronomic oral temozolomide as measured by 6 months overall survival (OS) after diagnosis of relapse or tumour progression in children and adolescents with relapsed or refractory high-grade malignant glioma and diffuse intrinsic pontine glioma.

Secondary objectives include:

1. To evaluate the safety and toxicity of the study treatment by common toxicity criteria (CTC; version 4.0).
2. To assess

   * the response rates at 6 months (continuous complete response = CCR, complete response = CR, partial response = PR, stable disease = SD, progressive disease = PD) and
   * progression-free survival (PFS) at 6 months, and
   * response rates, OS, and PFS at 12 months after relapse diagnosis or diagnosis of tumor progression. Response will be presented including histopathological variants.
3. To assess the pharmacokinetics of cilengitide administered as part of the study treatment.

Indication and study population for this trial:

Treatment of relapsed or refractory high grade gliomas and diffuse intrinsic pontine gliomas in paediatric patients ≥ 3 years and < 18 years of age.

Patients included in the study receive

* Cilengitide 1800 mg/m² i.v. twice weekly
* Temozolomide 75 mg/m²/d p.o. for 6 weeks, followed by 1 week rest with a mandatory platelet-count dependent dose adaptation rule: mandatory blood counts twice weekely: Platelets ≥ 100 000/µl (≥ 100 Gpt/l): 75 mg/m², platelets ≥ 50 000 - < 100 000/µl (≥ 50 - <100 Gpt/l): 50 mg/m², platelets < 50 000/µl (<50 Gpt/l): stop temozolomide until platelet recovery ≥ 100 000/µl (≥100 Gpt/l)
* Study treatment in the individual patient is scheduled for 1 year unless tumor progression or excessive toxicity occurs. However, study treatment may be extended beyond 1 year upon individual decision.

DETAILED DESCRIPTION:
Indication:

Treatment of relapsed or refractory high grade gliomas and diffuse intrinsic pontine gliomas in paediatric patients ≥ 3 years and < 18 years of age.

Background and rationale:

Relapsed or refractory high-grade gliomas or diffuse intrinsic pontine gliomas (in the following both addressed as high grade gliomas = HGG) in children and adolescents represent a very bad prognosis group for which a recommended standard salvage therapy is currently not available.

The combination of cilengitide and metronomic temozolomide will be investigated in the present trial as new treatment strategy for these patients.

Metronomic temozolomide was shown to act via inhibition of tumour angiogenesis and as a cytotoxic agent. Cilengitide might act via tumour angiogenesis and also inhibits tumour cell migration.

For both drugs, safe doses with only low toxicity had been defined in phase I trials for paediatric patients with recurrent or refractory brain tumours (Cilengitide: 1800 mg/m² twice weekly; metronomic Temozolomide: 75-80 mg/m²/d in a 6 week schedule followed by one week rest) In a phase II trial for adult patients with relapsed glioblastoma cilengitide as single agent showed a trend towards higher efficacy with 2000 mg twice weekly as compared to 500 mg twice weekly. Furthermore, in a phase II trial of newly diagnosed adult glioblastoma patients, signs of clinical activity of cilengitide in combination with radiotherapy and conventional temozolomide was seen in the methylated MGMT gene promoter subgroup. Based on these findings, a large randomized phase III trial investigating cilengitide in combination with standard therapy (temozolomide and radiation) in this subgroup was started recently.

Metronomic temozolomide was also shown to be still effective in glioma patients suffering from relapse after temozolomide standard therapy. Interestingly, the mode of action appears to be widely independent of the MGMT status, probably due to MGMT depletion by continuous treatment.

In conclusion, for both drugs signs of clinical activity have been shown in relapsed glioblastoma patients, even after failure of temozolomide standard therapy.

Study design:

Prospective, non-randomized phase II trial.

Study population:

Patients 3 years and < 18 years of age with high grade glioma or diffuse intrinsic pontine glioma relapsed after or refractory to standard therapy recruited by approved trial sites

Sample size:

It is planned to include 33 patients.

Therapy:

Patients included in the study receive

* Cilengitide 1800 mg/m² i.v. twice weekly
* Temozolomide 75 mg/m²/d p.o. for 6 weeks, followed by 1 week rest with a mandatory platelet-count dependent dose adaptation rule: mandatory blood counts twice weekely: Platelets ≥ 100 000/µl (≥ 100 Gpt/l): 75 mg/m², platelets ≥ 50 000 - < 100 000/µl (≥ 50 - <100 Gpt/l): 50 mg/m², platelets < 50 000/µl (<50 Gpt/l): stop temozolomide until platelet recovery ≥ 100 000/µl (≥100 Gpt/l)
* Study treatment in the individual patient is scheduled for 1 year unless tumor progression or excessive toxicity occurs. However, study treatment may be extended beyond 1 year upon individual decision.

Biometry:

Statistical analysis and sample size calculation:

The feasibility and efficacy of the HIT-HGG-CilMetro therapy will be assessed by a single stage analysis. Sample size calculation is based on the 6 month overall survival rate. This survival rate was found to be 44% in a historical study population from the HIT-GBM data base. An overall survival rate of 59% in the present study is considered to be of clinical relevance. Based on a one sided one sample χ2-test and a significance level α=5% a sample size of 33 patients is planned. This sample size implies a power of 50%.

Schedule:

The study is scheduled to start on January 1, 2012. The recruitment period for the trial will last 24 months until December 31, 2013. Individual follow-up for at least 1 year after study entry is required for this protocol. The study will be finished 30 days after completion of study treatment of the last patient enrolled, i.e. the expected end of the trial will be January 31, 2015.

Long-term follow-up is strongly recommended and will be organised via the HIT-HGG Study Office.

If the start of the study is delayed, given dates will change accordingly.

Financial support:

Merck KGaA, Darmstadt, Germany, provides a grant for the conduct of the trial, supplies Cilengitide free of charge and agrees to perform the laboratory assessments for pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of high-grade malignant glioma confirmed by central neuropathological review (last MRI diagnosis not older than 4 weeks) - including glioblastoma multiforme (WHO IV), anaplastic astrocytoma (WHO III), anaplastic oligodendroglioma (WHO III), anaplastic oligoastrocytoma (WHO III), anaplastic pilocytic astrocytoma (WHO III), anaplastic ganglioglioma (WHO III), anaplastic pleomorphic xanthoastrocytoma (analogous to WHO III), giant cell glioblastoma (WHO IV), and gliosarcoma (WHO IV) - or diagnosis of diffuse intrinsic pontine glioma confirmed by central neuroradiological review - refractory to standard treatment, or relapsed or progressive after first-line therapy.
2. Patient aged 3 years and older but under 18 years at time of relapse diagnosis
3. Written informed consent of the patient (mandatory from 15 years of age) or the parents (mandatory till 18 years of age).

Exclusion Criteria:

1. Known hypersensitivity or contraindication to any study drugs
2. Other (simultaneous) malignancies
3. Pregnancy and / or lactation
4. Patients who are sexually active refusing to use effective contraception (oral contraception, intrauterine devices, barrier method of contraception in conjunction with spermicidal jelly or surgical sterile)
5. Current or recent (within 30 days prior to start of trial treatment) treatment with another investigational drug or participation in another investigational trial
6. Severe concomitant diseases (e.g. immune deficiency syndrome) or HIV infection
7. Severe psychological disease or neurological damage without possibility to communicate
8. Clinical signs of intracranial pressure
9. Intracerebral hemorrhage or history of intracerebral hemorrhage
10. Requirements for laboratory test results not older than 2 weeks before patient´s inclusion:

    Platelets < 100 000/µl (< 100 Gpt/l) PT, INR and PTT above normal range Absulute neutrophil count ≤ 1 500/µl (< 1,5 Gpt/l) Hemoglobin < 10g/dl (< 6,4 mmol/L) Serum creatinine ≥ 1,5 x upper limit of normal range or creatinine clearance rate ≤ 60 ml/min/m2 (corrected for body surface area) Total bilirubin ≥ 1,5 x upper limit of normal range SGOT (ASAT) and SGPT (ALAT) ≥ 2,5 x upper limit of normal range Alkaline phosphatase ≥ 2,5 x upper limit of normal range
11. Hereditary Intrinsic Platelet Disorders
12. Ongoing irradiation or chemotherapy (within the last 4 weeks)
13. Estimated life expectancy of less than 2 months

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of a combined treatment with cilengitide and temozolomide as measured by 6 months overall survival after diagnosis of relapsed or refractory high grade glioma or diffuse intrinsic pontine glioma in children and adolescents | 6 months
  Evaluation of overall survival after 6 months

SECONDARY OUTCOMES:
Safety and toxicity of the study treatment | Up to 52 weeks of treatment and subsequently 30 days after end of treatment
  Evaluation of safety and toxicity of the study treatment by NCI Common Toxicity Criteria (CTC; version 4.0) for up to 30 days after the end of study treatment which may last up to 52 weeks.
  Toxic events defined as CTC grade 4 toxicities and deaths caused by therapy (CTC grade 5) excluding haematological toxicities (CTC grade 1-4)will be immediately assessed after documentation, and probability for such a toxic event statistically evaluated to ensure that this probability is within the predefined range (p1=15%).
Response rates (RR) at 6 months, progression-free survival (PFS) at 6 months, and RR, overall survival (OS), and PFS at 12 months after relapse diagnosis or diagnosis of tumor progression | Response rates and progression-free survival at 6 and 12 months, overall survival at 12 months (Trial subjects will be followed up for at least 1 year and 30 days after study entry)
  Evaluation of RR (continuous complete response = CCR, complete response = CR, partial response = PR, stable disease = SD, progressive disease = PD) by MRI and PFS (defined as survival from date of first progression/relapse to first documented date of second progression/relapse) after 6 and 12 months.
  Evaluation of OS after 12 months
Peak plasma levels of cilengitide [ng/ml] on day 1 of week 1 and day 4 of week 6 | Day 1 of treatment week 1: Immediately before and immediately after as well as 2, 4, and 7 hours after end of cilengitide administration; day 4 of treatment week 6: 2 hours after end of cilengitide adminstration
  Assessment of cilengitide serum levels [ng/ml] by a validated liquid chromatograpy tandem mass spectrometry assay on day 1 of week (before, immediately after, and 2, 4, 7 hours after cilengitide administration) and day 4 of week 6 (2 hours after cilengitide administration)

CONTACTS AND LOCATIONS:
Overall Officials: Christof M. Kramm, MD, Study Chair — University Children´s Hospital, Halle, Germany
Locations (1):
- University Children´s Hospital, Halle, Saxony-Anhalt, Germany